CLINICAL TRIAL: NCT06684912
Title: Acute Effects of Moderate Intensity Continuous Exercise Versus High-Intensity Interval Exercise on Flow Mediated Slowing and Flow Mediated Dilation in Adults with and Without Type 2 Diabetes
Brief Title: Acute Effects of Aerobic Exercise on Flow Mediated Slowing and Flow Mediated Dilation in Adults with and Without Type 2 Diabetes
Acronym: ARM WRESTLING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ARM WRESTLING
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: acute exercise; aerobic exercise; high intensity aerobic exercise; moderate continuous aerobic training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CONTROL (No Intervention): A non-exercise condition.
- High intensity interval exercise (HIIE) (Experimental): The HIIE was comprised of 1 min exercise bouts at 90% of oxygen uptake (V̇O2) reserve interspersed by 1 min active recovery bouts at 60% V̇O2 reserve (1:1).
  Interventions: Other: High-intensity interval exercise
- Moderate-intensity exercise (MICE) (Experimental): MICE at 60% V̇O2 reserve with the duration adjusted to each participant so that each participant achieved the target energy expenditure.
  Interventions: Other: Moderate continuous exercise

INTERVENTIONS:
Other: High-intensity interval exercise — The number of bouts of exercise-recovery for each participant was tailored to achieve the desired EE. For example, a participant with a peak oxygen uptake (V̇O2) peak of 30 mL.kg-1.min-1, weighing 80 kg, would need 6 bouts to match the target EE, assuming 1L of O2 uptake equals 5 kcal.
  Arms: High intensity interval exercise (HIIE)
Other: Moderate continuous exercise — Energy expenditure of exercise conditions (HIIE and MICE) were matched for energy expenditure. A participant with a V̇O2 peak of 30 mL.kg-1.min-1, weighing 80 kg, would need 6 bouts to match the target EE, assuming 1L of O2 uptake equals 5 kcal.
  Other Names: MICE
  Arms: Moderate-intensity exercise (MICE)

SUMMARY:
The endothelium is a protective lining of cells inside blood vessels. It keeps blood vessels working smoothly by controlling how wide or narrow your blood vessels are and protecting them from damage. Normally, the endothelium keeps a healthy balance between signals that relax or tighten blood vessels. But with advancing age or certain diseases like diabetes, this balance is disrupted. This can make blood vessels weaker and lead to serious problems in the heart and other organs.

Researchers use a test called brachial flow-mediated dilation (FMD) to check how well blood vessels work. FMD shows how good blood vessels are at making a chemical called nitric oxide (NO), which helps them relax and widen. During the FMD test, researchers reduce blood flow for a short time with a blood pressure cuff, then release it to see how blood vessels respond. They use an ultrasound machine to measure this. While FMD is useful, it has some downsides-it's hard to do right, needs expensive tools, and experts don't always agree on how to analyze the results. A newer method called flow-mediated slowing (FMS) aims to fix these problems. FMS uses pulse wave velocity (PWV) to measure how stiff your blood vessels are. Stiffer vessels mean less nitric oxide and a higher chance of heart problems. After reducing blood flow with a blood pressure cuff and releasing it, healthy people show a drop in PWV (reduction in arterial stiffness), but people with heart failure or high blood pressure do not. Thus, FMS holds promise as it is an easier way to measure blood vessel health.

Exercise training helps keep blood vessels healthy with advancing age. Research has shown that regular aerobic exercise, (running or biking), and strength exercise (lifting weights), can improve how blood vessels work and make them less stiff. This is true even for healthy people. For people with type 2 diabetes, exercise training is even more important to preserve blood vessel health. The intensity of exercise may determine how much blood vessels improve. Research has shown that high-intensity interval training (HIIT)-where you switch between hard exercise and rest-works better than steady, moderate exercise for making blood vessels healthier and less stiff. It is thought that HIIT improves blood vessel health partly by improving how the body uses insulin. Still, not all studies show that training improves blood vessel health in people with type 2 diabetes.

A single session of exercise presents a challenge to blood vessels that allows researchers to understand how exercise over time improves blood vessel health. In addition, studying how blood vessels react to one workout (called the acute exercise model) is helpful because researchers can easily control things like the type of exercise, how hard it is, or how long it lasts. Acute exercise research also helps control other factors, such as nutrition, that may bias results. Thus, acute exercise research is a great method to learn how exercise works in the short term and how it might help in the long run.

Therefore, the present study aimed to determine how FMD and FMS respond after an acute bout of high-intensity interval exercise and moderate continuous exercise in older adults without type 2 diabetes, and also healthy young adults.

The key research questions were:

1. Is the FMD and FMS response after an acute bout of exercise dependent on exercise intensity?
2. Is the FMD and FMS response after an acute bout of exercise dependent on age and disease status?

All participants were asked to:

Complete two exercise sessions - one moderate- and one high-intensity interval bout on a treadmill. The order of the sessions was randomly assigned, similar to flipping a coin.

FMD and FMS were measured before and after each acute exercise bout in the laboratory.

The researchers compared FMD and FMS responses between exercise intensities (high vs. moderate) and populations (individuals with and without type diabetes).

DETAILED DESCRIPTION:
The study was designed as a randomized, cross-over, repeated-measures experiment. Participants attended 3 separate intervention sessions consisting of an acute bout of HIIE, an acute bout of MICE, or a no exercise (CON) condition, in randomized order (http://www.randomizer.org/) to which participants were blinded until arrival at the laboratory. On a separate day before the interventions, all participants performed a cardiopulmonary exercise test (CPET). The exercise sessions began and ended with a warm-up and a cool-down, respectively, with a duration of 3 min each at 60% of V̇O2 reserve. Both the HIIE and MICE protocols were designed to match a weekly energy expenditure (EE) of 8 kcal.kg-1 week-1 comprising 3 hypothetical exercise sessions per week. Both protocols were individually tailored to each participant regarding his weight and peak oxygen uptake (V̇O2 peak), and the prescribed target intensities were supervised by an exercise physiologist with a heart rate monitor (Garmin, US) throughout the session. To eliminate the possible diurnal variation, each participant performed all interventions at an equal time of day (in the mornings) with a minimum of 48h between sessions. Post-exercise measurements at 10 and 60 min were aimed to characterize the post-exercise biphasic response of the brachial endothelial function. Participants reported to the laboratory in a fasting state (≥ 4h) and refrained from vigorous exercise, vitamin supplements, foods/drinks containing caffeine, and alcohol for at least 24h before each session.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 30 kg/m2
* Less than two risk factors for cardiovascular disease (for participants without type diabetes mellitus)
* No electrocardiographic or symptomatic abnormalities on the exercise stress
* Physically active (3-5 days of structured exercise; for participants without type diabetes)
* Glycosylated haemoglobin (HbA1c) levels (≥ 5.7% and bellow 8.0%) or fasting blood glucose ≥126 mg/dL and below 185 mg/dL) - for participants with type 2 diabetes

Exclusion Criteria:

* Cardiovascular disease (e.g., heart failure, ischemic heart disease)
* Orthostatic intolerance
* Thyroid dysfunction
* Mental disease
* Microvascular complications (e.g., neuropathies)
* Renal disease
* Musculoskeletal disease (e.g., sarcopenia, osteoporosis)
* Smoking
* Vasoactive medications (e.g. angiotensin-converting enzyme inhibitors, calcium channel blockers)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Brachial endothelial function | Before and 10, and 60-minutes after acute aerobic exercise
  Brachial artery flow-mediated dilation - ultrasound
Brachial artery stiffness | Before and 5, and 60-minutes after acute aerobic exercise
  Brachial artery flow-mediated slowing - ultrasound

SECONDARY OUTCOMES:
Central arterial stiffness | Before and 10, and 60-minutes after acute aerobic exercise
  Applanation tonometry - carotid-femoral pulse wave velocity
Upper limb arterial stiffness | Before and 10, and 60-minutes after acute aerobic exercise
  Applanation tonometry - carotid-radial pulse wave velocity
Lower limb arterial stiffness | Before and 10, and 60-minutes after acute aerobic exercise
  Applanation tonometry - carotid-dorsalis pedis pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Melo, PhD, Principal Investigator — Egas Moniz School of Health & Science
Locations (1):
- Faculdade de Motricidade Humana - University of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with an academic interest in vascular responses to exercise in people with type 2 diabetes. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Background] Francois ME, Little JP. The impact of acute high-intensity interval exercise on biomarkers of cardiovascular health in type 2 diabetes. Eur J Appl Physiol. 2017 Aug;117(8):1607-1616. doi: 10.1007/s00421-017-3649-2. Epub 2017 May 31. PMID 28567668
- [Background] Magalhaes JP, Melo X, Correia IR, Ribeiro RT, Raposo J, Dores H, Bicho M, Sardinha LB. Effects of combined training with different intensities on vascular health in patients with type 2 diabetes: a 1-year randomized controlled trial. Cardiovasc Diabetol. 2019 Mar 18;18(1):34. doi: 10.1186/s12933-019-0840-2. PMID 30885194
- [Background] Colberg SR, Albright AL, Blissmer BJ, Braun B, Chasan-Taber L, Fernhall B, Regensteiner JG, Rubin RR, Sigal RJ; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: American College of Sports Medicine and the American Diabetes Association: joint position statement. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2010 Dec;42(12):2282-303. doi: 10.1249/MSS.0b013e3181eeb61c. PMID 21084931
- [Background] Fiuza-Luces C, Santos-Lozano A, Joyner M, Carrera-Bastos P, Picazo O, Zugaza JL, Izquierdo M, Ruilope LM, Lucia A. Exercise benefits in cardiovascular disease: beyond attenuation of traditional risk factors. Nat Rev Cardiol. 2018 Dec;15(12):731-743. doi: 10.1038/s41569-018-0065-1. PMID 30115967
- [Background] Ashor AW, Lara J, Siervo M, Celis-Morales C, Oggioni C, Jakovljevic DG, Mathers JC. Exercise modalities and endothelial function: a systematic review and dose-response meta-analysis of randomized controlled trials. Sports Med. 2015 Feb;45(2):279-96. doi: 10.1007/s40279-014-0272-9. PMID 25281334
- [Background] Ellins EA, New KJ, Datta DB, Watkins S, Haralambos K, Rees A, Aled Rees D, Halcox JP. Validation of a new method for non-invasive assessment of vasomotor function. Eur J Prev Cardiol. 2016 Apr;23(6):577-83. doi: 10.1177/2047487315597210. Epub 2015 Jul 24. PMID 26209709
- [Background] Naka KK, Tweddel AC, Doshi SN, Goodfellow J, Henderson AH. Flow-mediated changes in pulse wave velocity: a new clinical measure of endothelial function. Eur Heart J. 2006 Feb;27(3):302-9. doi: 10.1093/eurheartj/ehi619. Epub 2005 Nov 2. PMID 16267075
- [Background] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Background] Cahill PA, Redmond EM. Vascular endothelium - Gatekeeper of vessel health. Atherosclerosis. 2016 May;248:97-109. doi: 10.1016/j.atherosclerosis.2016.03.007. Epub 2016 Mar 9. PMID 26994427